CLINICAL TRIAL: NCT00530075
Title: Phase II Study on Gusperimus in Patients With Refractory Wegener's Granulomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nippon Kayaku Co., Ltd. (Industry)
Responsible Party: Peter A. Heinzel, Ph.D., Clinical and Scientific Department, Euro Nippon Kayaku GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2007-09

CONDITIONS: Wegener's Granulomatosis
Keywords: Wegener Granulomatosis; Vasculitis; Gusperimus; Immunosuppression
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Vasculitis | interventions — gusperimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Gusperimus
  Interventions: Drug: Gusperimus

INTERVENTIONS:
Drug: Gusperimus — SC, 0.5mg/kg/day, consecutive 21 days administration, 1 to 2 weeks rest, 6 cycles

SUMMARY:
Wegener's granulomatosis is a primary systemic vasculitis characterized by granulomatous and necrotizing inflammation predominantly affecting the respiratory tract and the kidneys. Conventional therapy of Wegener's granulomatosis with cyclophosphamide and corticosteroids is limited by incomplete remissions and a high relapse rate. Patients accumulate irreversible damage due to the disease and the consequences of prolonged drug exposure. The efficacy and safety of an alternative immunosuppressive drug, gusperimus, was evaluated in patients with refractory disease. A prospective, international, nulti-centre, single limb, open label study. Entry required active Wegener's granulomatosis with a Birmingham Vasculitis Activity Score (BVAS) >=4 and previous therapy with cyclophosphamide or methotrexate. Immunosuppressive drugs were withdrawn at entry and prednisolone doses adjusted according to clinical status. Gusperimus, 0.5mg/kg/day, was self-administered by subcutaneous injection in six treatment cycles of 21 days with a seven day washout between cycles. Cycles were stopped early for white blood count < 4,000/mm3. The primary endpoint was complete remission (BVAS=0 for at least 2 months) or partial remission (BVAS<50% of entry score). After the sixth cycle azathioprine was commenced and follow-up continued for a further six months.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of WG according to American College of Rheumatology (ACR) and Chapel Hill Consensus Conference (CHCC) definition
* BVAS >= 4
* Total disease duration >= 3 months treated with CYC or >= 6 months with MTX
* Age 18 - 80
* WBC >= 4,000/mm3, haemoglobin >= 8g/dl, neutrophils >= 2,500/mm3, platelets >= 100,000/mm3
* ALT, bilirubin and alkaline phosphatase levels within 2x the upper limits of normal
* Documented to be non-pregnant by serum/urine pregnancy test
* Willing to participate in this study
* Provide signed informed consent
* Able and prepared to self-administer the study drug or have a close friend/relative able to do this

Exclusion Criteria:

* Participation in another clinical research study
* Pregnant or nursing mothers and women of childbearing age not using appropriate contraception
* Clear evidence of active disease due to bacteria/viral infection
* Patient has an unacceptable risk for participation in a study of immunosuppressive therapy
* History of substance abuse or psychotic disorders
* Previous treatment with Gusperimus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-12; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jayne, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (7):
- General Faculty Hospital, Prague, Czechia
- Reumatologisk Klinik, Copenhagen, Denmark
- Universitatsklinikum Schleswig-Holstein, Lübeck, Germany
- University Hospital Maastricht, Maastricht, Netherlands
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (2):
  - Western General Hospital, Edinburgh, Scotland
  - Addenbrookes Hospital, Cambridge

REFERENCES:
- [Background] Birck R, Warnatz K, Lorenz HM, Choi M, Haubitz M, Grunke M, Peter HH, Kalden JR, Gobel U, Drexler JM, Hotta O, Nowack R, Van Der Woude FJ. 15-Deoxyspergualin in patients with refractory ANCA-associated systemic vasculitis: a six-month open-label trial to evaluate safety and efficacy. J Am Soc Nephrol. 2003 Feb;14(2):440-7. doi: 10.1097/01.asn.0000048716.42876.14. PMID 12538745
- See also: The European Vasculitis Study Group — http://www.vasculitis.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 sites in 6 European countries from 2003 to 2006
Groups:
- Gusperimus: SC, 0.5mg/kg/day, consecutive 21 days administration, 7 days rest, 6 cycles
Period: Overall Study
Arm/Group | Gusperimus
Started | 45
Completed | 38
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Lack of Efficacy | 3
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gusperimus
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: Years] | 51 [19 to 77]
Gender [Count of Participants; unit: Participants]
  Female | 16
  Male | 29
Region of Enrollment [Number; unit: participants]
  Europe | 45

OUTCOME MEASURES:

1. Primary Outcome: Remission of Vasculitis
Description: The primary efficacy outcome measure was remission of vasculitis. Complete remission was defined as a Birmingham vasculitis activity score (BVAS) of 0 sustained for at least 2 months. Partial remission was defined as a reduction in BVAS of 50% or more, sustained for at least 2 months, when compared with the BVAS at entry.
  Entry required active Wegener's granulomatosis with a BVAS >= 4. Their disease had to be active, as measured with BVAS in which clinical manifestations caused by active vasculitis are scored on a list of predefined organ-specific items.
Time Frame: At Entry (Day 1 of Cycle 1), Day 22 of cycles 1-6, up to 24 weeks
Population: Efficacy Population
Measure: Number; unit: Percentage of participants
Arm/Group | Gusperimus
Number analyzed (Participants) | 44
Percentage of participants | 95

2. Secondary Outcome: Duration of Clinical Response
Description: Time from Complete Remission or Partial Remission to Relapse.
Time Frame: At Entry (Day 1 of Cycle 1), Day 22 of cycles 1-6, up to 24 weeks, End of treatment period, and 3 and 6 months of follow-up period
Population: Patients who had relapsed after achieved at least partial remission
Measure: Median (Full Range); unit: Days
Arm/Group | Gusperimus
Number analyzed (Participants) | 18
Days | 170 [44 to 316]

3. Secondary Outcome: Haematuria
Description: Assessment of anti-inflammatory activity of gusperimus using surrogate marker: number of hematuria-positive patients.
Time Frame: At Entry (Day 1 of Cycle 1), End of treatment period, up to 24 weeks
Population: Efficacy population
Measure: Number; unit: Number of participants
Arm/Group | Gusperimus
Number analyzed (Participants) | 44
Number of participants
  At Entry | 16
  End of treatment period | 6

4. Secondary Outcome: Creatinine
Description: Assessment of anti-inflammatory activity of gusperimus using surrogate marker: serum creatinine level
Time Frame: At Entry (Day 1 of Cycle 1), End of treatment period, up to 24 weeks
Population: Efficacy population
Measure: Median (Full Range); unit: micromol/L
Arm/Group | Gusperimus
Number analyzed (Participants) | 44
micromol/L
  At Entry | 130 [58 to 299]
  End of treatment period | 132 [72 to 279]

5. Secondary Outcome: ANCA
Description: Assessment of anti-neutrophil cytoplasmic antibody (ANCA): Number of ANCA-positive patients was counted.
  ANCA are highly associatred with active WG, with c-ANCA titres observed in 90% of WG. In addition to their diagnostic value, it has been suggested that ANCA may have a predictive value for relapse in patients with systemic vasculitis.
Time Frame: At Entry (Day 1 of Cycle 1), End of treatment period, up to 24 weeks
Population: Efficacy Population
Measure: Number; unit: Number of participants
Arm/Group | Gusperimus
Number analyzed (Participants) | 44
Number of participants
  At Entry | 39
  End of treatment period | 34

6. Secondary Outcome: CRP
Description: Assessment of anti-inflammatory activity of gusperimus using surrogate marker: serum C-reactive protein level.
Time Frame: At Entry (Day 1 of Cycle 1), End of treatment period, up to 24 weeks
Population: Patients who had elevated CRP level (> 6 mg/dL) at entry
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Gusperimus
Number analyzed (Participants) | 23
mg/dL
  At Entry | 17.5 [7 to 88]
  End of treatment period | 9 [1 to 124]

7. Secondary Outcome: Vasculitis Damage Index (VDI)
Description: Assessment of the degree of irreversible damage due to the vasculitis using VDI scoring system. The VDI comprises 64 items of damage (grouped into 11 organ-based systems). Total VDI score is 0 - 64. The higher scores represent the more severe damage occurred in patients. The VDI score can either increase or remain the same over time.
Time Frame: At Entry (Day 1 of Cycle 1), End of treatment period, up to 24 weeks, 6 months of follow-up period
Population: Efficacy Population
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Gusperimus
Number analyzed (Participants) | 44
Score on a scale
  At Entry | 4.5 [0 to 14]
  End of treatment period | 5 [0 to 16]
  6 months of follow-up period | 5 [0 to 16]

8. Secondary Outcome: SF-36
Description: Assessment of the impact of gusperimus on general health using the Short form-36 (SF-36) questionaire. The SF-36 is a self-report, 36 item survey measuring health-related quality-of-life. Thirty-five items are used to construct 8 scales: (1) physical functioning, (2) role physical, (3) bodily pain, (4) general health, (5) vitality, (6) social function, (7) role emotional, and (8) mental health. Raw scores are calculated as the sum of re-coded scale items and transformed to a 0 to 100 scale. If scores for all 8 scales are available, two summary measures known as component scores are derived: the Physical Health Component Score (PCS) and the Mental Health Component Score (MCS). First each scale standardized to the relevant population. Then PCS and MCS are calculated as the weighted sum of standardized scores. All scales and the component scores are positively scored so that higher scores represent better health-related quality-of-life.
Time Frame: At Entry (Day 1 of Cycle 1), End of treatment period, up to 24 weeks
Population: Efficacy Population
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Gusperimus
Number analyzed (Participants) | 44
Score on a scale
  Physical component score (at Entry) | 29.6 [14.8 to 50.2]
  Physical component score (at End of treatment peri | 34.3 [11.6 to 53.7]
  Mental component score (at Entry) | 49.4 [21.0 to 62.9]
  Mental component score (at End of treatment period | 48 [23.7 to 62.8]

ADVERSE EVENTS:
Time Frame: Throughout study period, up to 24 weeks
Arm/Group | Gusperimus
Serious Adverse Events (participants affected / at risk) | 17/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gusperimus (N=45)
Leucopaenia/Anaemia (Blood and lymphatic system disorders) | 7
Infections (Infections and infestations) | 7
Bronchopneumonia (Infections and infestations) | 5
Dental abscess (Infections and infestations) | 1
Campylobacter jejuni diarrhoea (Infections and infestations) | 1
Relapses of Wegener's granulomatosis (Respiratory, thoracic and mediastinal disorders) | 4
Acute upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 2
Active Wegener's granulomatosis (Respiratory, thoracic and mediastinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gusperimus (N=45)
Anaemia (Blood and lymphatic system disorders) | 8
Leucopaenia (Blood and lymphatic system disorders) | 17
Lower respiratory tract infection (Infections and infestations) | 12
Upper respiratory tract infection (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 6
Candida infection (Infections and infestations) | 7
Injection site pain/pruritus (General disorders) | 26
Injection site haemorrhage (General disorders) | 8
Pain oral cavity/throat (Gastrointestinal disorders) | 19
Dysgeusia (Nervous system disorders) | 8
Stomatitis/mouth ulcers (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 16
Vomoting (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 8
Acne (Skin and subcutaneous tissue disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No